CLINICAL TRIAL: NCT01129843
Title: A Cluster Randomized Trial for Lowering Prevalence of Anemia in Rural Hilly Villages With Directly Observed Home Based Daily Iron Therapy(DOHBIT)
Brief Title: Directly Observed Iron Supplementation to Treat Anemia
Acronym: DOHBIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Build Healthy India Movement (Other)
Collaborators: Ministry of Science and Technology, India (Other Government)
Responsible Party: Dr Sahul Bharti, Build Healthy India Movement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No.SSD/WS/102/2008
Record Dates: First submitted 2010-05-22; First posted 2010-05-25 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Iron Deficiency Anemia (IDA)
Keywords: anemia; iron deficiency; nutritional; iron supplementation; cluster randomized control trial
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia; Iron Deficiencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Directly observed home based daily iron therapy (Experimental): Village volunteers will provide directly observed home based daily iron supplementation( ferrous sulphate) to enrolled anemic women in the experimental arm
  Interventions: Drug: Directly observed home based daily iron therapy
- Clinic driven unsupervised daily iron therapy (Active Comparator): In the control group of villages, clinic driven unsupervised iron ( ferrous sulphate) supplementation will be offered on monthly basis to anemic women for 3 months
  Interventions: Drug: Directly observed home based daily iron therapy

INTERVENTIONS:
Drug: Directly observed home based daily iron therapy — Directly Observed Home based Daily Iron( ferrous sulphate) therapy (DOHBIT) will be provided to the anemic women by the local village volunteers. Dose of elemental iron therapy will be 100 mg once daily for mild to moderate anemia and twice daily for severe anemia for a cumulative duration of 90 days

SUMMARY:
India continues to be one of the countries with very high prevalence of anemia. In fact, National Family Health Survey-3 (NFHS-3,2005-06) revealed increasing prevalence of anemia in women and children, since NFHS-2 in 1998-99. In the backdrop of this alarming trend, the aim of this trial is to assess the effectiveness of a community based anemia management intervention ( curative and holistic) delivered to rural anemia women and girls(aged 13 years and above)in remote hilly villages (unit of randomization) in terms of change in anemia prevalence (unit of analysis) after 3 months of iron supplementation. This trial with a therapeutic component of "Directly Observed Home Based daily Iron Therapy (DOHBIT)" by local village volunteers is conceived as a whole community approach to improve the hemoglobin status of affected patients in remote villages.

DETAILED DESCRIPTION:
To combat iron deficiency anemia, the challenge is not so much knowing "what" to do, but to understand "how" to implement effective and sustainable interventions. In this perspective, the aim of this trial is to assess the effectiveness of a community based anemia management therapeutic intervention delivered to rural anemic women (aged 13 years and above) in remote hilly villages (unit of randomization) in terms of change in anemia prevalence (unit of analysis) after 3 months of iron supplementation.

The intervention programme "Directly Observed Home Based daily Iron Therapy"(DOHBIT) by local village volunteers is conceived as a whole community approach to improve the hemoglobin status of affected patients in remote villages. A cluster-randomized trial will be thus the design of choice from the outset. For intervention arm of trial, each anemic patient will receive DOHBIT (Directly Observed Home Based daily Iron Therapy) by local village volunteer for a total of 90 days whereas in the control arm of trial each patient will receive usual standard iron therapy without daily supervision for the same duration. Information, educational and counseling strategies will be similar for the two groups.

Primary outcome will be the anemia prevalence (difference of proportions) in intervention vs. control groups after trial intervention. Secondary outcomes in two groups include mean hemoglobin levels, compliance and side effects of iron therapy, body mass index and quality of life scores.

Sample size estimates, adjusted for cluster randomization (assuming Intracluster Correlation Coefficient of 0.05 and mean cluster size of 30 patients/village based on our pilot study), show that with 10 villages, each for intervention and control groups, an average 300 anemic patients per treatment arm would need to be treated to provide sufficient power to determine a 20% difference in anemia prevalence in two groups- a reduction deemed to a worthwhile impact of the intervention to be reliably detected at 80% power.

Then a statistically valid approach to the analysis of primary outcome variable will be to calculate a single outcome measure for each randomized unit and apply standard parametric method (chi-square) to the set of summary measures, keeping in mind that any conclusion will be strictly applicable only at the cluster level. Since, covariate adjustment will be required on an individual level for various secondary outcomes, thus a different approach based on the individual, as unit of analysis, adjusting for clustering will be more appropriate in analyzing various secondary outcome measures.

Overall, DOHBIT is one of the strategies to increase the capacity of individuals and communities to define, analyze and act to address their own health needs. Moreover, in the supply-demand continuum, DOHBIT by utilizing facilitators and motivators at the local level will optimize demand as well as supply of iron supplementation programme in the community.

ELIGIBILITY:
Inclusion Criteria:

* Women and adolescent girls aged 13 years and above who are diagnosed with anemia using WHO defined cut-offs for hemoglobin levels

Exclusion Criteria:

* Any active medical disease ( acute or chronic)other than anemia, any subject already on iron supplementation for >4 weeks, any subject with significant mental impairment, recent history of Gastrointestinal bleed

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of anemia | 1 year
  Compare the prevalence of anemia in two cluster randomized groups of villages

SECONDARY OUTCOMES:
Compliance with iron therapy | 1 year
  To compare the degree of compliance with iron therapy by anemic women between two cluster randomized groups of villages

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sahul Bharti, MD Pediatrics, PDCC, Dip Stats, Principal Investigator — Build Healthy India Movement (BHIM)
Locations (1):
- Build Healthy India Movement, Sirmaur, Himachal Pradesh, India

REFERENCES:
- [Background] Bharti S. Feasibility of "directly observed home-based twice-daily iron therapy" (DOHBIT) for management of anemia in rural patients: a pilot study. Indian J Med Sci. 2004 Oct;58(10):431-8. PMID 15523164